CLINICAL TRIAL: NCT05420025
Title: THE EFFECT OF VIRTUAL REALITY GLASSES APPLICATION ON PAIN ANXIETY FEAR AND PHYSIOLOGICAL PARAMETERS OCCURING DURING DRESSING CHANGE IN CHILDREN WITH LIVER TRANSPLANT
Brief Title: VIRTUAL REALITY GLASSES, CHILDREN WITH LIVER TRANSPLANTATION
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Semiha Dertli, Research Assistant, Firat University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Firat Universityyyyyyyyyyy; Emine ERDEM (Other: ERCIYES UNIVERSITY); Tevfik Tolga SAHIN (Other: INONU UNIVERSITY)
Record Dates: First submitted 2022-06-11; First posted 2022-06-15 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Children With Liver Transplant
Keywords: Liver transplantation; Virtual Reality; Pain; Anxiety; Fear; Dressing chang; Child
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Quasi Experimental
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CHILDREN APPLIED WITH VIRTUAL REALITY GLASSES (Experimental): Before the first dressing (5 minutes before the dressing) of the children who were accepted to the Organ Transplantation A Service from the intensive care unit after the transplantation, the introductory characteristics form and scales will be applied and the physiological parameters of the child (heart rate, respiratory rate, blood pressure) will be applied by the researcher. , oxygen saturation) will be taken. Then the children will be put on SGG and the glasses will be synchronized. During the dressing, children will be shown a video with SGG, which received expert opinion beforehand. After the dressing, the physiological parameters of the children will be measured again and the scales will be applied again.

INTERVENTIONS:
Other:

SUMMARY:
The aim of the study is to determine the effect of SGG application on pain, anxiety/anxiety, fear and physiological variables during dressing in children aged 4-10 years with liver transplantation.

Children with liver transplantation are in the whole treatment and care process; exposed to frequent and repetitive painful procedures. Abdominal dressings were observed to be the most frequent-repetitive, long-term source of pain affecting children physically and psychologically from these procedures. It is thought that the use of virtual reality during abdominal dressing will be beneficial because of the size of the abdominal incision and dressings, the use of no analgesic or sedative agent during dressing, and the children are affected by this incision image. It is thought that virtual reality can be used and effective in this area in terms of keeping people away from images and sounds and isolating them from real life.

DETAILED DESCRIPTION:
Liver transplantation is becoming widespread as an effective treatment option. Medical and technological developments have affected the increase in the number and success rate of transplant patients. On the other hand, some physiological and psychological problems occur in children during and after transplantation. It is stated that the biggest source of fear for children in the hospital is invasive procedures such as blood draw, injection, and post-operative dressing change. These interventions, which are accepted as treatment and care procedures and which must be performed, are defined as procedural sources of pain. Dressing changes after abdominal surgery can cause the child to experience pain and fear. Although it is known that procedural pain is physiological, it is thought that the fear and anxiety that arise during this time also cause pain. The pain experienced by children during dressing change and the inability to effectively manage this pain; It can disrupt the secretion of hormones and permanently change the function and arrangement of some organs. It can prolong hospital stay by causing deterioration in glucose balance and delay in wound healing. Procedural pain management aims to minimize the pain and anxiety experienced by children due to medical interventions. For this purpose, it is recommended to use non-pharmacological methods in addition to pharmacological treatment methods. One of the most preferred non-pharmacological methods in children is distraction. Unlike other methods of distraction, virtual reality is a different method in that it distances the person from images and sounds, isolates them from real life, brings together multiple sensory experiences and maximizes the sense of attention. In the treatment and care process of children with liver transplantation; exposed to frequent and repetitive painful procedures. Abdominal dressings were observed to be the most frequent-repetitive, long-term source of pain affecting children physically and psychologically from these procedures. It is thought that the use of virtual reality during abdominal dressing will be beneficial because of the size of the abdominal incision and dressings, the use of an analgesic/sedative agent during dressing, and the fact that children are affected by this incision image.

The aim of the study was to determine the effect of SGG application on pain, anxiety/anxiety, fear and physiological variables during dressing in children aged 4-10 years who had liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 4-10,
* do not have a chronic or genetic disease,
* not mentally, visually or hearing impaired,
* no painful intervention is applied at least one hour before the dressing,
* no analgesic and sedative applied at least one hour before the dressing,
* both himself and his parents are open to communication and cooperation,
* Children who are first dressed in the service, who both themselves and their parents volunteer to participate in the study, and who give verbal and written consent will be included.

Exclusion Criteria:

- Children who cannot adapt to the virtual reality glasses during the study, who are restless and who want to withdraw from the study will be excluded from the study.

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2022-04-26 (Actual); Primary Completion 2023-02-25 (Estimated); Study Completion 2023-05-27 (Estimated)

PRIMARY OUTCOMES:
Faces Pain Scale-Revised (FPSR) | 5- 10 min
  Hicks et al. (2001) Revised Facial Expressions Pain Scale (R-FAS) is a self-expression-based scale that can be applied to children aged 4-16. The scale consists of 6 facial expressions graded from 0 to 10 according to the severity of the pain. The R-FLPS, which can be understood easily and quickly with the explanation given to children, has been translated into more than 35 languages. Values between 1-3 indicate mild pain, values between 4-6 indicate moderate pain, and values between 7-10 indicate severe pain.
Child Anxiety Scale-State Scale (CAS-D) | 5-10 min
  CAS-D is a visual scale for children aged 4-10 years. With a light bulb at the bottom and ten horizontal lines running towards the top, this visual scale resembles a thermometer. While applying the scale; children "Imagine that all of your anxious or nervous feelings are on the bulb or the top of the thermometer (point with your finger on the scale)", "If you are even slightly worried or nervous, the emotions may increase a little (point your finger up on the scale)", "Very, very worried or If you are nervous, the emotions may go all the way to the top of the lines (move your finger to the top), instructions such as "Put a line to let us know how anxious or nervous you are feeling." Following the data collection process, the research team members followed the child's "ÇAS-D " and a transparent meter with ½ point increments is placed over the child's rating and the ½ point increment is rounded to the nearest number to determine the child's score. The score can range from 0-10.
Child Fear Scale (CFS) | 5-10 Min
  The Child Fear Scale (CDS), developed by McMurtry et al., is used to evaluate the fear levels of children aged 4-10 (32). 5 cartoon face images were used in the scale. Anxiety level is evaluated with numbers between "0" and "4". A score of "0" indicates "no anxiety" and a score of "4" indicates "severe anxiety". Validity and reliability of the scale Özalp-Geker et al. Made by in 2018. The scope validity index is 0.89.

CONTACTS AND LOCATIONS:
Locations (1):
- Firat University, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No